CLINICAL TRIAL: NCT05918627
Title: A Randomized, Double-blind, Placebo-controlled, Dose Escalating Study to Examine the Safety, Tolerability and Pharmacokinetic Profile of Single Oral Doses of SLx-2119 in Healthy Male Subjects
Brief Title: A Study to Determine the Effect of Multiple Oral Doses of SLx-2119 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kadmon, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: SLx-2119-09-01; U1111-1291-6021 (Other: ICTRP)
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Immune System Disorder (Healthy Volunteer)
MeSH Terms: conditions — Immune System Diseases | interventions — KD025

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Dose level 1 (Experimental): Single Oral Doses of 20 mg SLx-2119 or placebo on Day 1
  Interventions: Drug: Belumosudil mesylate; Drug: Placebo
- Dose level 2 (Experimental): Single Oral Doses of 40 mg SLx-2119 or placebo on Day 1
  Interventions: Drug: Belumosudil mesylate; Drug: Placebo
- Dose level 3 (Experimental): Single Oral Doses of 80 mg SLx-2119 or placebo on Day 1
  Interventions: Drug: Belumosudil mesylate; Drug: Placebo
- Dose level 4 (Experimental): Single Oral Doses of 160 mg SLx-2119 or placebo on Day 1
  Interventions: Drug: Belumosudil mesylate; Drug: Placebo
- Dose level 5 (Experimental): Single Oral Doses of 320 mg SLx-2119 or placebo on Day 1
  Interventions: Drug: Belumosudil mesylate; Drug: Placebo
- Dose level 6 (Experimental): Single Oral Doses of 640 mg SLx-2119 or placebo on Day 1
  Interventions: Drug: Belumosudil mesylate; Drug: Placebo

INTERVENTIONS:
Drug: Belumosudil mesylate — Pharmaceutical form: capsule; Route of administration: oral
  Other Names: SLx-2119; KD025; SAR445761
Drug: Placebo — Pharmaceutical form: capsule; Route of administration: oral

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and pharmacokinetics of multiple doses of SLx-2119 in healthy male participants.

DETAILED DESCRIPTION:
Duration per participants is Day 1 up to 30 days after participant is treated with the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants between the ages of 18 and 55 years, inclusive.
* Able to provide written informed consent prior to the performance of any study specific procedures.
* Body mass index (BMI) range of 19-30 kilogram per square meter (kg/m2), inclusive.

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:
* Past or present disease that is judged by the investigator to have the potential to interfere with the study procedures, compromise safety, or affect the PK evaluations.
* Known sensitivity to Rho-associated coiled-coil containing serine/threonine protein kinases (ROCK2) inhibitor agents or to any of the constituents of the KD025 formulation.

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-09-21 (Actual); Primary Completion 2009-12-09 (Actual); Study Completion 2009-12-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events and serious adverse events | Day 1 up to approximately 30 days after participant is treated with the last dose of study drug.
  Safety observations and measurements include AEs, safety laboratory tests, vital sign measurements, physical examinations, and ECGs.

SECONDARY OUTCOMES:
Cmax of SLx-2119 and its metabolites (SLx-2131 and SLx-3047) | Predose and multiple timepoints up to 24 hours postdose on Day 1
  Cmax is maximum plasma concentration determined directly from the concentration time profile
tmax of SLx-2119 and its metabolites (SLx-2131 and SLx-3047) | Predose and multiple timepoints up to 24 hours postdose on Day 1
  tmax is observed time to reach peak plasma concentration
AUC0-24 of SLx-2119 and its metabolites (SLx-2131 and SLx-3047) | Predose and multiple timepoints up to 24 hours postdose on Day 1
  AUC0-24 is area under the plasma concentration-time curve from predose (time 0) to 24 hours Postdose
AUCinf of SLx-2119 and its metabolites (SLx-2131 and SLx-3047) | Predose and multiple timepoints up to 24 hours postdose on Day 1
  AUCinf is area under the concentration-time curve from predose (time 0) extrapolated to Infinity
t1/2 of SLx-2119 and its metabolites (SLx-2131 and SLx-3047) | Predose and multiple timepoints up to 24 hours postdose on Day 1
  t1/2 is terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org